CLINICAL TRIAL: NCT04805164
Title: Evaluation of the Efficiency of the Bone Substitute Cerament-G Locally Delivering Gentamicin in the Treatment of Chronic Osteomyelitis of Long Bones: Randomized Multicentre Study in the CRIOAc Network - CONVICTION Study
Brief Title: Evaluation of the Efficiency of the Bone Substitute Cerament-G Locally Delivering Gentamicin in the Treatment of Chronic Osteomyelitis of Long Bones
Acronym: CONVICTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL20_0065; 2020-A02299-30 (Other: ANSM)
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Osteomyelitis Chronic
Keywords: Bone infection; chronic osteomyelitis; bone substitute

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovative strategy (Experimental): usual medical and surgical care with corticotomy and use of a bone substitute (Cerament-G) delivering gentamicin locally (± skin and soft-tissue/muscle flap) and antibiotic therapy.
  Interventions: Procedure: Corticotomy and use of the bone substitute : Cerament-G device.
- Reference strategy (Active Comparator): Medico-surgical usual care with corticotomy (± skin and soft-tissue/muscle flap), and antibiotic therapy.
  Interventions: Procedure: Corticotomy

INTERVENTIONS:
Procedure: Corticotomy and use of the bone substitute : Cerament-G device. — Corticotomy and Cerament-G device
  Arms: Innovative strategy
Procedure: Corticotomy — Corticotomy
  Arms: Reference strategy

SUMMARY:
Chronic osteomyelitis is a serious osteoarticular infection that most often occurs in the long bones (tibia, femur, humerus), responsible for significant morbidity with risk of fracture and amputation. It is due to the presence of bacteria in the bone marrow, sometimes responsible for an intraosseous abscess.

Chronic osteomyelitis can have a hematogenous or more often exogenous origin, after trauma or surgery. The bacteria involved have the ability to modify their metabolism and involve persistence mechanisms (such as biofilm) making them difficult to eradicate. The treatment of chronic osteomyelitis requires surgery, i.e. corticotomy, which means opening of the bone cortex to perform an endomedullary curettage to identify the bacteria, remove any sequestration (bone fragments to which the bacteria adhere as biofilm) and reduce the bacterial inoculum. At the same time, or at a second stage, a skin and soft tissue/muscle flap may be required, especially in patients with long-standing disease with embrittlement and adhesion of the skin and soft tissue to the underlying bone.

Post-operatively, the patient receives a probabilistic systemic antibiotic therapy and then a systemic antibiotic therapy targeted on the identified germ, for a period of 3 months. The effectiveness of these antibiotics is based on their ability to penetrate bone tissue. Despite the progress made in both antibiotics and surgical treatments, the probability of failure (recurrence of infection) is around 20%, and has unfortunately remained stable for more than 20 years.

Cerament-G (BONESUPPORT AB Laboratory, Sweden), a synthetic bone substitute composed of hydroxyapatite, calcium sulphate, and gentamicin, fills the "dead space" formed during surgery, prevents infection of this blood-filled cavity, and promotes bone regeneration within this space (limiting the risk of fracture in the medium and long term). Cerament-G also delivers locally very high doses of gentamicin (concentration of 17.5 mg/mL in the device) for several weeks. Gentamicine is a broad-spectrum bactericidal antibiotic effective against the vast majority of bacteria involved in osteoarticular infections. It provides effective local antibiotic therapy through wide exposure and prolonged concentrations during several weeks.

To date, there is no other bone substitute with antibiotics available in France. Two prospective studies have shown that Cerament-G reduces the number of infectious recurrences (about 5%).

This innovation is available in France but at a high price (between 2,500 and 4,000 euros) and is not currently reimbursed. However, the use of this product would make it possible to improve the health and quality of life of patients while avoiding certain consumption of resources.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected chronic osteomyelitis (stage III of the Cierny-Mader classification) of a long bone of the tibia, femur, humerus or forearm, at the diaphysis, metaphysis or epiphysis, defined as follows:

  * Supposed inoculation > 3 months ;
  * At least one of the following clinical signs at the suspected infected site:

    * Spontaneous or supporting pain ;
    * Presence of fistula; or history of fistula discharge
    * Presence of serous or purulent flow;
    * Presence of bone exposure;
    * Local Inflammation;
    * Fever in the absence of any other explanation.
  * At least one of the following radiological signs at the suspected infected site:

    * Bone reshaping with osteolysis or periosteal apposition;
    * Presence of intramedullary abscess (if MRI performed);
    * Presence of a fistulous pathway to the intramedullary (if MRI performed);
    * Presence of bone sequestration visible on CT scan (if CT scan performed).
* Patient in whom conventional surgical treatment of chronic osteomyelitis is possible, with decortication and corticotomy with endomedullary curettage (to eradicate bone sequestrums, reduce the inoculum, and identify the bacterium(s) involved) and secondary intramedullary residual cavity;
* Patient in whom 3 months of systemic antibiotic therapy post-operatively are planned;
* If osteosynthetic material is present in the infection site, this material should be considered preoperatively as completely removable during chronic osteomyelitis surgery;
* Patient in whom a direct closure without tension is possible, or in whom a skin and soft-tissue/muscle flap can be performed within 15 days after the initial surgery;
* Male or female patient between 18 and 80 years of age;
* Patient who has given written informed consent to participate in the study;
* Geographically stable patient;
* Patient able to comply with follow-up visits, protocol schedule and therapeutic treatment, according to investigator's judgement;
* Affiliated patient or beneficiary of a social security system

Exclusion Criteria:

* Acute hematogenic osteomyelitis (Cierny-Mader stage I) ;
* Cortical osteitis (Cierny-Mader stage II);
* Septic pseudoarthrosis (Cierny-Mader stage IV);
* Patient requiring an estimated skin and soft-tissue/muscle flap that cannot be done within 15 days after surgery for the treatment of chronic osteomyelitis;
* Woman who is pregnant, nursing or who is considering becoming pregnant during the study period;
* Patient participating in another interventional study that could interfere with it;
* Patient known to have hypersensitivity to aminoglycosides (especially gentamicin), sulfites (including calcium sulfate) or calcium hydroxyapatite;
* Contraindication to the use of Cerament-G: severe myasthenia (class IV or higher according to the MGFA classification), , severe renal insufficiency (creatinine clearance <30 mL/min according to the Cockcroft-Gault formula, or GFR < 30 ml/min/1.73² according to the CKD-EPI or MDRDs equation or, dialysis patient), pre-existing disorders of calcium metabolism (total plasma calcium (or total corrected plasma calcium according to albuminemia) outside normal laboratory values);
* Patient with endocrine or metabolic disorders known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, hyperthyroidism, parathyroid disorder, Ehler-Danlos syndrome, osteogenesis imperfecta);
* Patient with one or more untreated malignant cancers (including Marjolin's ulcer), or undergoing radiotherapy or chemotherapy;
* Adult patient protected by law, under guardianship or trusteeship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2027-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Utility Ratio (ICUR) between the two treatments strategies for chronic long bone osteomyelitis | At 24 months (M24)

SECONDARY OUTCOMES:
Recurrence of bone infection | At 24 months (M24)
  Proportion of patients with at least one recurrence of infection on the studied bone and time to recurrence. The Event Validation Committee will confirm the recurrence of infection.
Intraoperative and Postoperative complications | From inclusion to 24 months (M24)
  Number and types of intraoperative and postoperative complications up to 24 months (including fracture) according to CTCAE and Clavien-Dindo classifications; and proportion of patients with at least one complication during follow-up
Repeated surgeries for complication | From first surgery to 24 months (M24)
  Number of repeat surgeries for complication up to 24 months; and proportion of patients who had at least one repeat surgery for complication during follow-up
Proportion of patients with amputations | At 24 months (M24)
  Proportion of patients with amputation of the area containing the bone studied.
Bone healing and bone remodelling/consolidation | At 12 months (M12)
  Proportion of patients with bone healing and proportion of patients with bone remodelling/consolidation, assessed from a standard radiograph (confirmed by the Event Validation Committee).
Serious Adverse Events (SAEs) attributable to systemic antibiotic therapy. | Within 3 months of the first intervention (M3)
  Number and types of serious adverse events (SAEs) attributable to systemic antibiotic therapy following the first intervention; and proportion of patients with at least one SAE attributable to this systemic antibiotic therapy; within 3 months of the first intervention.
Acute renal failure | Within 3 months of the first procedure (M3)
  Proportion of patients with acute renal failure within 3 months of the first procedure
Adverse Events related to the use of Cerament-G | At 24 months (M24)
  Cost of both strategies estimated at 24 months
Real cost | 24 months (M24)
  Real cost associated of a corticotomy procedure using Cerament-G
Estimated utility | At inclusion, at Week 4/Week 6, Month 3, Month 6, Month12, Month 18 and Month 24 (usual follow-up visits) as well as after each repeat surgery according to the same schedule
  Estimated utility measured with the EQ-5D (EuroQol Group-5 dimensions) questionnaire.
Estimated incremental cost-effectiveness ratio | At 24 months (M24)
  Estimated incremental cost-effectiveness ratio with no recurrence of infection as efficacy endpoint
Budgetary impact analysis | 24 months (M24)
  Budgetary impact analysis carried out from the perspective of the French Health Insurance.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Amiens-Picardie, Amiens
  - CHU de Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - APHP, Boulogne-Billancourt
  - CHU Brest, Brest
  - CHU de Caen, Caen
  - CHU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHRU Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de Toulouse, Toulouse